CLINICAL TRIAL: NCT06517628
Title: The Heart Outcomes in Pregnancy Expectations for Mom and Baby Study
Acronym: HOPE
Status: Recruiting | Type: Observational
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: Albert Einstein College of Medicine (Other); Baylor College of Medicine (Other); Beth Israel Deaconess Medical Center, Inc. (Unknown); The Children's Hospital Corporation (Unknown); The Brigham and Women's Hospital, Inc. (Unknown); The Trustees of Columbia University in the City of New York (Unknown); Henry Ford Hospital (Other); The Johns Hopkins University (Unknown); The Miriam Hospital/Lifespan (Unknown); The General Hospital Corporation d/b/a Massachusetts General Hospital (Unknown); Northwell Health (Other); Northwestern University (Other); Oregon Health and Science University (Other); Saint Luke's Health System Inc. (Unknown); Board of Trustees of the Leland Stanford Junior University (Unknown); The Research Foundation for the State University of New York (Unknown); The Regents of the University of California, Irvine (Unknown); The Regents of the University of California, Los Angeles (Unknown); University of North Carolina, Chapel Hill (Other); The Board of Trustees of the University of Illinois (Unknown); Trustees of Indiana University (Unknown); University of Kansas Medical Center (Other); University of Massachusetts Chan Medical School (Unknown); Regents of the University of Michigan (Unknown); University of Mississippi Medical Center (Other); The Curators of the University of Missouri (Unknown); The Trustees of the University of Pennsylvania (Unknown); University of Pittsburgh (Other); The University of South Florida Board of Trustees for University of South Florida (Unknown); University of Washington (Other); University of Texas Southwestern Medical Center (Other); Weil Medical Colleqe of Cornell University (Unknown); Women and Infants Hospital of Rhode Island (Other); Tennessee Maternal Fetal Medicine PLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0073599
Record Dates: First submitted 2024-07-08; First posted 2024-07-24 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy Complications, Cardiovascular
Keywords: Pregnancy, cardio-obstetrics; Structures of Care; Quality of Care; Disparities; Heart disease in pregnancy; Pregnancy complications; Adverse pregnancy outcomes; Major adverse cardiac events; Neonatal adverse events; Quality of life
MeSH Terms: conditions — Pregnancy Complications, Cardiovascular; Pregnancy Complications; Cardiovascular Diseases | interventions — Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant people with cardiovascular disease: Any pregnant patient with acquired or congenital cardiovascular disease upon presentation to a cardio-obstetrics clinic.
  Interventions: Other: Purely observational study on the care and outcomes of participants with cardiovascular disease in pregnancy.

INTERVENTIONS:
Other: Purely observational study on the care and outcomes of participants with cardiovascular disease in pregnancy. — The primary exposure variable is the organization of cardio-obstetrics care which will be defined by annual site surveys and its association with outcomes will be defined by hierarchical models adjusting for patient characteristics.

SUMMARY:
This is a prospective, observational study which is evaluating the obstetrical, neonatal, and cardiovascular outcomes of 1000 pregnant people with known heart disease to define how best to structure cardio-obstetrics care to optimize outcomes.

DETAILED DESCRIPTION:
The US is the only industrialized nation to experience a rise in maternal mortality over the last decade. Despite the Healthy People 2030 agenda target of reducing maternal mortality by 10%, rates in the United States are predicted to increase. Furthermore, maternal mortality disproportionately impacts Black, Hispanic, American Indian/Alaskan Native (AIAN), and Asian/Pacific Islander birthing people, who die at a rate that far greater than their White counterparts. Black birthing people are twice as likely to experience severe maternal morbidity (SMM) and 3-4X more likely to die, even after adjusting for demographic and hospital factors. Unfortunately, this gap is widening, with a 20% increase in death for Blacks as compared with a 5% rise in Whites over the last decade. Understanding contributors to adverse outcomes for marginalized birthing populations cannot solely be determined from retrospective chart adjudication and requires prospective evaluation to better understand patient and treatment factors contributing to maternal morbidity and mortality.

Despite affecting only 2-4% of pregnancies, cardiovascular disease (CVD) accounts for >30% of maternal deaths, making it a leading cause of maternal mortality for all birthing people and the number one cause in the Black population. Pregnant people with acquired and congenital heart disease experience the majority of CV-related morbidity and mortality, of which over three quarters have been deemed preventable. The prevalence of CVD is expected to grow as risk factors for CV-related death (obesity, advanced maternal age, hypertensive disorders, and preexisting heart disease) are rising dramatically in pregnant people, which disproportionately burdens marginalized populations. Provider-based factors are a leading cause of preventable morbidity, yet the lack of evidence-based guidelines, means of risk-stratifying pregnant people with CVD, or insight into how best to structure care limits the ability to improve maternal outcomes.

Mortality is not the only important outcome for pregnant people with CVD. For every maternal death, it is estimated that 100 people - 50,000 per year - will suffer severe maternal morbidity (SMM) during delivery, with significant costs to both their families and the economy. Adverse pregnancy outcomes (APOs) and neonatal adverse clinical events (NACEs), including pre-eclampsia, preterm delivery, fetal growth restriction, stillbirth and maternal hemorrhage, are all significantly more common in those with heart disease. Pregnant people who survive these events are more likely to suffer post-traumatic stress and depression, which can adversely impact mother-child bonding and long-term health. Importantly, there are no studies in this population evaluating quality of life, which cannot be measured using retrospective data.

To address the critical need for reversing the US trend in maternal morbidity and mortality, the Heart Outcomes in Pregnancy Expectations (HOPE) study will focus on the highest risk population, pregnant people with CVD. It will provide deeper insights into maternal risk factors, their association with care, and the influence of alternative structures of cardio-obstetric care with APO, MACE, and NACE outcomes. It is a multi-site, multidisciplinary prospective study at >30 cardio-obstetrics clinics throughout the US with a key secondary goal of better understanding racial disparities in care and outcomes. Not only will traditional APOs, MACE, and NACE events from presentation to 1-year after delivery be collected, generic and disease-specific quality of life will be measured as a way to evaluate their independent impact on outcomes.

Preliminary insights through our pilot program highlight the importance of better structures of care as a means of improving outcomes, which has previously been established in other clinical settings, but not in cardio-obstetrics care. The investigators have identified 6 key structures of care that have been variably adopted through the US and for which additional data to define their independent association with outcomes is needed.

These include:

1. multidisciplinary (OB/maternal-fetal medicine [MFM], cardiology, anesthesia, critical care, etc.) care teams;
2. a COB care coordinator;
3. coordinated inter-disciplinary patient evaluation;
4. team debriefing
5. the ability to perform high-risk deliveries in the ICU and
6. formalized warm hand offs to primary or sub-specialty care after delivery.

After adjusting for extensive patient factors associated with adverse outcomes, the independent association of these structures of care with outcomes will be estimated as a foundation for testing and disseminating those that are most effective.

ELIGIBILITY:
Inclusion:

Must have one or more condition(s) within the 6 following categories - Repaired or Unrepaired

* Congenital or structural heart disease
* Aortopathies
* Arrhythmias
* Cardiomyopathies and Heart Failure
* Coronary disease
* Other (Current endocarditis or history of endocarditis, Pericarditis, Pericardial effusion - Moderate or Large, Pericardial constriction, Pulmonary hypertension (all types) defined as mean pulmonary artery systolic pressure of >20 mmHg by right heart catheterization or pulmonary hypertension estimated in the severe range by echo)

Exclusion Criteria

* Unable to participate in telephone follow-up
* Too hard of hearing to do follow-up by telephone or deaf
* Incarcerated prisoner
* History of dementia.
* Subjects without a way for contact by telephone for follow-up
* Refused participation in the study
* Unable to consent for self
* Traumatic Aortic Disease
* Peripartum cardiomyopathy diagnosed in current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant people with cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Adverse pregnancy outcomes | up to 6 weeks postpartum
  HELLP, preeclampsia, gestational hypertension, eclampsia, superimposed preeclampsia on chronic hypertension (SIPE), premature preterm rupture of membranes (PPROM), preterm delivery, thrombotic complications, hemorrhage, maternal mortality, placental abruption, Admission ICU delivery

SECONDARY OUTCOMES:
Rate of Maternal Adverse Cardiac Events (MACE) | Up to 1 year postpartum
  A composite outcome including any of the following: cardiovascular death, non-fatal stroke, myocardial infarction, hospitalization for acute coronary syndromes, urgent revascularization procedures, decompensated heart failure, aortic dissection, clinically significant arrhythmia requiring treatment (eg. atrial fibrillation/flutter, SVT, ventricular tachycardia, etc), cardiac transplant
Rate of Neonatal adverse clinical events (NACE) | Through maternal hospital discharge
  A composite outcome including any of the following: APGARS < 8 at 5 minutes, birthweight of < 2500 grams, NICU admission, supplemental oxygen use, neonatal death, fetal death, spontaneous abortion/miscarriage, intrauterine fetal growth restriction

OTHER OUTCOMES:
Changes in Generic Quality of Life as Assessed by the Short Form-36 | Through 1 year post partum
  All patients will complete the Short Form-36 on enrollment and changes over time through 1 year after delivery and will be compared by patient characteristics and structures of care.
Changes in Depressive Symptoms, as Assessed by the Edinburgh Postpartum Depression Scale | Through 1 year post partum
  This questionnaire will be completed on enrollment and changes over time through 1 year after delivery and will be compared by patient characteristics and structures of care.
Experiences with pregnancy care and delivery will be assessed with the Childbirth Experience Survey | Third trimester and 6 weeks after delivery
  This questionnaire will be completed during the 3rd trimester and 6 weeks after delivery and will be compared by patient characteristics and structures of care.
Perceived Discrimination will be assessed using the Experience of Depression Scale | Enrollment and 6 and 12 months after delivery
  This questionnaire will be completed on enrollment and at 6 and 12 months after delivery so that cross-sectional and changes over time through 1 year after delivery can be compared by patient characteristics and structures of care.
Self-perceived Health Status will be assessed using a version of the Kansas City Cardiomyopathy Questionnaire Modified for Pregnancy | Enrollment, 3rd Trimester, and 6 weeks, 6 months and 12 months after delivery
  This questionnaire will be completed on enrollment and changes over time through 1 year after delivery will be compared by patient characteristics and structures of care.
Coronary-specific Health Status over Time among Participants with a History of Coronary Disease | Enrollment, 3rd Trimester, and 6 weeks and 12 months after delivery
  This questionnaire will be completed by participants with a history of coronary artery disease (including SCAD) on enrollment and changes over time through 1 year after delivery and will be compared by patient characteristics and structures of care.
Atrial Fibrillation-specific Health Status over Time among Participants with a History of Atrial Fibrillation | Enrollment, 3rd Trimester, and 6 weeks and 12 months after delivery
  This questionnaire will be completed by participants with a history of atrial fibrillation on enrollment and changes over time through 1 year after delivery and will be compared by patient characteristics and structures of care.
Disease-specific Health Status over Time among Participants with a History of Congenital Heart Disease | Enrollment, 3rd Trimester, and 6 weeks and 12 months after delivery
  This questionnaire will be completed by participants with a history of congenital heart disease on enrollment and changes over time through 1 year after delivery and will be compared by patient characteristics and structures of care.

CONTACTS AND LOCATIONS:
Overall Officials: John Spertus, MD, MPH, Principal Investigator — University of Missouri, Kansas City
Locations (1):
- Saint Luke's Hospital of Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited into BioLincc (https://biolincc.nhlbi.nih.gov/). These data will be provided in a completely de-identified format with random shifting of dates that are internally consistent with the participant's actual experiences.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The HOPE team commits to providing the data as soon as possible, but no sooner than 1 year after the completion of follow-up of the last patient. The Steering/Publications Committee will annually review any additions to the data set, including the creation of composite variables, to explore whether updates to the deposited data are needed and, if so, these will be made within 3 months of their creation/addition.
Access Criteria: unrestricted